CLINICAL TRIAL: NCT04110210
Title: Effectiveness of Bilateral Ultrasound-Guided Erector Spinae Plane Block in Intraoperative and Postoperative Pain Control in Lumbar Spine Surgeries.A Randomized Controlled Trial
Brief Title: Effectiveness of Bilateral Ultrasound-Guided Erector Spinae Plane Block
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abdalla, Professor of Anesthesia &I.C.U and Pain Clinic, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: MD-80-2019
Record Dates: First submitted 2019-03-15; First posted 2019-10-01 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Erector Spinae Plane Block

STUDY DESIGN:
Intervention Model Description: Following skin sterilization and local anesthetic infiltration of the superficial tissues, an echogenic 22-G block needle is inserted in-plane to the ultrasound beam in a cranial-to-caudal direction until contact was made with the transverse process. Correct location of the needle tip in the fascial plane deep to erector spinae muscle is confirmed by injecting 0.5-1 ml saline and seeing the fluid lifting the erector spinae muscle off the transverse process while not distending the muscle. A total of 20ml bupivacaine 0.25% are then injected into the ESP. The procedure is repeated on the contralateral side.
Who Masked: Participant, Care Provider
Masking Description: Prospective randomized double blinded clinical study on humans
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A(Ultrasound guided ESP block after indtiucon of GA). (Active Comparator): Following skin sterilization and local anesthetic infiltration of the superficial tissues, an echogenic 22-G block needle is inserted in-plane to the ultrasound beam in a cranial-to-caudal direction until contact was made with the transverse process. Correct location of the needle tip in the fascial plane deep to erector spinae muscle is confirmed by injecting 0.5-1 ml saline and seeing the fluid lifting the erector spinae muscle off the transverse process while not distending the muscle. A total of 20ml bupivacaine 0.25% are then injected into the ESP. The procedure is repeated on the contralateral side.
  Interventions: Drug: Bilateral Ultrasound-Guided Erector Spinae Plane Block
- Group B(GA with conventional analgesia) (Active Comparator): After operation, patients will be transferred to post anesthesia care unit (PACU) for complete recovery and monitoring. The pain VAS scores between the studied groups will be registered every 4 hours for 24 hours postoperatively. A standard postoperative analgesia regimen will be prescribed as paracetamol 1gm every 6 hours and ketorolac 30mg every 8 hours in the first 24 hours postoperatively. Morphine 2.5 mg will be given as a rescue analgesic dose if visual analogue score was ≥ 3 or when patient suffering from pain between the assessment intervals in both groups not exceeding 0.1 mg/kg in a period of 6 hours. Metoclopramide 0.15 mg/kg IV will be prescribed for patients complaining of nausea or vomiting.
  Interventions: Drug: Morphine Consumption

INTERVENTIONS:
Drug: Bilateral Ultrasound-Guided Erector Spinae Plane Block — Following skin sterilization and local anesthetic infiltration of the superficial tissues, an echogenic 22-G block needle is inserted in-plane to the ultrasound beam in a cranial-to-caudal direction until contact was made with the transverse process. Correct location of the needle tip in the fascial plane deep to erector spinae muscle is confirmed by injecting 0.5-1 ml saline and seeing the fluid lifting the erector spinae muscle off the transverse process while not distending the muscle. A total of 20ml bupivacaine 0.25% are then injected into the ESP. The procedure is repeated on the contralateral side.
  Arms: Group A(Ultrasound guided ESP block after indtiucon of GA).
Drug: Morphine Consumption — After operation, patients will be transferred to post anesthesia care unit (PACU) for complete recovery and monitoring. The pain VAS scores between the studied groups will be registered every 4 hours for 24 hours postoperatively. A standard postoperative analgesia regimen will be prescribed as paracetamol 1gm every 6 hours and ketorolac 30mg every 8 hours in the first 24 hours postoperatively. Morphine 2.5 mg will be given as a rescue analgesic dose if visual analogue score was ≥ 3 or when patient suffering from pain between the assessment intervals in both groups not exceeding 0.1 mg/kg in a period of 6 hours. Metoclopramide 0.15 mg/kg IV will be prescribed for patients complaining of nausea or vomiting.
  Arms: Group B(GA with conventional analgesia)

SUMMARY:
The proposed mechanism of action of the ESPB is via blockade of the dorsal and ventral rami of the spinal nerves and sympathetic nerve fibers. Radiographic evidence suggests that local anesthetic injected into at the ESP spreads both cranially and caudally as the plane is continuous along the vertebral column . ESPB reportshave demonstrated analgesia at cervical, thoracic, and lumbar levels for procedures such aspyeloplasty, lipoma excision, breast reconstruction,malignant mesothelioma, inguinal hernia repairs, and hip reconstructions

DETAILED DESCRIPTION:
One of these local analgesia is the erector spinae plane block (ESPB). it was first described in 2016 as a regional block for the treatment of thoracic neuropathic pain. This has shown promise as an alternative to neuraxial blockade for a variety of surgeries with good effect. In addition, the block has a reduced risk of epidural hematoma, direct spinal cord injury, and central infection .

The proposed mechanism of action of the ESPB is via blockade of the dorsal and ventral rami of the spinal nerves and sympathetic nerve fibers. Radiographic evidence suggests that local anesthetic injected into at the ESP spreads both cranially and caudally as the plane is continuous along the vertebral column . ESPB reportshave demonstrated analgesia at cervical, thoracic, and lumbar levels for procedures such aspyeloplasty, lipoma excision, breast reconstruction,malignant mesothelioma, inguinal hernia repairs, and hip reconstructions

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 to 60 years.
* Genders eligible for study: both sexes.
* ASA I-II.
* Undergoing lumbar spine surgeries in any 2 levels(L1-L5).
* BMI from 18.5 to 30 kg/m2

Exclusion Criteria:

* Patient refusal
* Contraindications to regional anesthesia (Bleeding disorders, Use of any anti-coagulants, local infection, etc.).
* Known allergy to local anesthetics.
* ASA III-IV.
* Patients aged less than 18 or more than 60.
* Body mass index >35.
* Patients with difficulty in evaluating their level of pain.
* Patients with secondary surgery or surgery involving more than two intervertebral spaces were excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2019-09-08 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Intraoperative and postoperative Opiate consumption | Up to 24 hours
  Intraoperative fentanyl and postoperative morphine consumption

SECONDARY OUTCOMES:
Time of the first postoperative analgesic request . | Up to 24 hours
  Time of the first postoperative analgesic request (duration of the block).
Visual Analouge score | Up to 24 hours
  Visual Analouge score score postoperative where 0=No Pain (better outcome) and 10=Intractable Pain (worse outcome)
Block onset | Up to 24 hours
  Onset of the block

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdalla Mohamed, M.D, Principal Investigator — Cairo University
Locations (1):
- Ahmed Abdalla Mohamed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Still Working